CLINICAL TRIAL: NCT06686394
Title: HERTHENA-Breast-01: A Phase 1b/2, Multicenter, Open-label, Dose-Finding Study to Evaluate the Safety and Antitumor Activity of Patritumab Deruxtecan in Participants With HER2 Positive Unresectable Locally Advanced Breast Cancer or Metastatic Breast Cancer
Brief Title: Study of Patritumab Deruxtecan With Other Anticancer Agents in Participants With HER2 Positive Breast Cancer That Has Spread and Cannot Be Surgically Removed (MK-1022-009)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1022-009; MK-1022-009 (Other: MSD); jRCT2041250022 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Breast Neoplasms; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — patritumab deruxtecan; Trastuzumab; Ogivri; Ontruzant; pertuzumab; tucatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Patritumab deruxtecan plus trastuzumab (Experimental): Participants receive patritumab deruxtecan intravenous (IV) infusion and trastuzumab or trastuzumab biosimilar IV infusion on Day 1 of each 21-day cycle (every 3 weeks) until disease progression, intolerable toxicity, or investigator decision.
  Interventions: Biological: Patritumab deruxtecan; Biological: Trastuzumab; Biological: Trastuzumab Biosimilar
- Patritumab deruxtecan plus pertuzumab and trastuzumab (Experimental): Participants receive patritumab deruxtecan IV infusion, pertuzumab IV infusion, and trastuzumab or trastuzumab biosimilar IV infusion on Day 1 of each 21-day cycle (every 3 weeks) until disease progression, intolerable toxicity, or investigator decision.
  Interventions: Biological: Patritumab deruxtecan; Biological: Trastuzumab; Biological: Trastuzumab Biosimilar; Biological: Pertuzumab
- Patritumab deruxtecan plus trastuzumab and tucatinib (Experimental): Participants receive patritumab deruxtecan IV infusion and trastuzumab or trastuzumab biosimilar IV infusion on Day 1 of each 21-day cycle (every 3 weeks), and tucatinib is administered orally twice daily for each 21-day cycle, until disease progression, intolerable toxicity, or investigator decision.
  Interventions: Biological: Patritumab deruxtecan; Biological: Trastuzumab; Biological: Trastuzumab Biosimilar; Biological: Tucatinib

INTERVENTIONS:
Biological: Patritumab deruxtecan — Patritumab deruxtecan administered via IV infusion
  Other Names: MK-1022; HER3-DXd; U3-1402
Biological: Trastuzumab — Trastuzumab administered via IV infusion
  Other Names: Herceptin®
Biological: Trastuzumab Biosimilar — Trastuzumab biosimilar administered via IV infusion
  Other Names: Trazimera®; Ogivri®; Herzuma®; Ontruzant®; Kanjinti®; Hercessi®
Biological: Pertuzumab — Pertuzumab administered via IV infusion
  Arms: Patritumab deruxtecan plus pertuzumab and trastuzumab
Biological: Tucatinib — Tucatinib administered as oral tablets
  Arms: Patritumab deruxtecan plus trastuzumab and tucatinib

SUMMARY:
Researchers want to learn if patritumab deruxtecan (MK-1022) can treat certain breast cancers. The breast cancers being studied are HER2 positive unresectable locally advanced or metastatic (the cancer has spread to other parts of the body). The goals of this study are to learn:

* About the safety and how well people tolerate of patritumab deruxtecan
* How many people have the cancer respond (get smaller or go away) to treatment

DETAILED DESCRIPTION:
The following countries will be participating in the trial: Canada, United Kingdom, Israel, Japan, South Korea, and USA.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has histologically confirmed HER2+ locally advanced unresectable breast cancer or metastatic breast cancer
* Human immunodeficiency virus (HIV)-infected participants must have well-controlled HIV on antiretroviral therapy (ART)
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received HBV antiviral therapy for at least 4 weeks, and have undetectable hepatitis B virus (HBV) viral load before allocation
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 within 7 days before start of study intervention

Arm 1:

* Has received at least a minimum of 2 and a maximum of 5 prior lines of anti-HER2 therapy in the locally advanced or metastatic setting
* Had disease progression on or after any previous trastuzumab deruxtecan (T-DXd) treatment

Arm 2:

-Has received no more than 5 prior lines of anti-HER2 therapy in the locally advanced or metastatic setting

Arm 3:

-Has received and had disease progression from T-DXd treatment in any setting and a maximum of 3 prior lines of anti-HER2 therapy in the locally advanced or metastatic setting. T-DXd must be the most recent therapy received before enrollment.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Uncontrolled or significant cardiovascular disease
* History of (noninfectious) pneumonitis/interstitial lung disease (ILD) that required steroids or has current pneumonitis/interstitial lung disease
* Has clinically severe respiratory compromise
* Has any history of or evidence of any current leptomeningeal disease
* Has clinically significant corneal disease
* Evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection
* HIV infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Known additional malignancy that is progressing or has required active treatment within the past 3 years
* Evidence of spinal cord compression or brain metastases
* Has an active infection requiring systemic therapy
* Concurrent active HBV and HCV infection
* Has had major surgical procedure (excluding placement of vascular access) less than 28 days

Arm 3 ONLY

- Has received prior treatment with tucatinib, lapatinib, or neratinib, or any investigational HER2-targeted tyrosine kinase inhibitors in the locally advanced or metastatic setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2030-04-18 (Estimated); Study Completion 2030-04-18 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-Limiting Toxicity (DLT) | Up to 21 days
  DLT will be defined as any drug-related AE observed during the DLT evaluation period that results in a change to a given dose or a delay in initiating the next cycle. The number of participants who experience a DLT will be presented.
Number of Participants with One or More Adverse Events (AEs) | Up to approximately 13 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who experience an AE will be presented.
Number of Participants who Discontinue Study Intervention Due to an AE | Up to approximately 12 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who discontinue study treatment due to an AE will be presented.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Patritumab Deruxtecan Antibody-Drug Conjugate (ADC) | At designated time points (up to ~13 months)
  Blood samples collected at designated time points will be used to determine the Cmax of patritumab deruxtecan ADC.
Trough Concentration (Ctrough) of Patritumab Deruxtecan ADC | At designated time points (up to ~13 months)
  Blood samples collected at designated time points will be used to determine the Ctrough of patritumab deruxtecan ADC.
Area Under the Plasma Concentration-Time Curve (AUC) of Patritumab Deruxtecan ADC | At designated time points (up to ~13 months)
  Blood samples collected at designated time points will be used to determine the AUC of patritumab deruxtecan ADC.
Maximum Plasma Concentration (Cmax) of Total Patritumab Deruxtecan Antidrug Antibody (ADA) | At designated time points (up to ~13 months)
  Blood samples collected at designated time points will be used to determine the Cmax of total patritumab deruxtecan ADA.
Trough Concentration (Ctrough) of Total Patritumab Deruxtecan ADA | At designated time points (up to ~13 months)
  Blood samples collected at designated time points will be used to determine the Ctrough of total patritumab deruxtecan ADA.
Area Under the Plasma Concentration-Time Curve (AUC) of Total Patritumab Deruxtecan ADA | At designated time points (up to ~13 months)
  Blood samples collected at designated time points will be used to determine the AUC of total patritumab deruxtecan ADA.
Maximum Plasma Concentration (Cmax) of Patritumab Deruxtecan Free Payload | At designated time points (up to ~13 months)
  Blood samples collected at designated time points will be used to determine the Cmax of patritumab deruxtecan free payload.
Trough Concentration (Ctrough) of Patritumab Deruxtecan Free Payload | At designated time points (up to ~13 months)
  Blood samples collected at designated time points will be used to determine the Ctrough of patritumab deruxtecan free payload.
Area Under the Plasma Concentration-Time Curve (AUC) of Patritumab Deruxtecan Free Payload | At designated time points (up to ~13 months)
  Blood samples collected at designated time points will be used to determine the AUC of patritumab deruxtecan free payload.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (16):
- United States (4):
  - Dana-Farber Cancer Institute ( Site 0050), Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey ( Site 0052), New Brunswick, New Jersey
  - Prisma Health - Upstate (ITOR)_Edenfield ( Site 0053), Greenville, South Carolina
  - Inova Schar Cancer Institute ( Site 0051), Fairfax, Virginia
- Canada (4):
  - Kingston General Hospital ( Site 0061), Kingston, Ontario
  - Princess Margaret Cancer Centre ( Site 0001), Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal ( Site 0004), Montreal, Quebec
  - Jewish General Hospital ( Site 0003), Montreal, Quebec
- Israel (3):
  - Rambam Health Care Campus ( Site 0011), Haifa
  - Rabin Medical Center ( Site 0012), Petah Tikva
  - Sheba Medical Center ( Site 0010), Ramat Gan
- Nagoya City University Hospital ( Site 0020), Nagoya, Aichi-ken, Japan
- South Korea (2):
  - Seoul National University Hospital ( Site 0030), Seoul
  - Asan Medical Center ( Site 0031), Seoul
- United Kingdom (2):
  - University College London Hospital ( Site 0041), London, Camden
  - St Bartholomew s Hospital ( Site 0040), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com